CLINICAL TRIAL: NCT01742910
Title: Posterior Capsule Opacification and Frequency of Nd:YAG Treatment and of Two Microincision IOLs: Tecnis ZCB00 and Acrysof SA60AT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Prof. Dr. Rupert Menapace, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: EK128/2008
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Capsule Opacification; Pseudophakia; Cataract
MeSH Terms: conditions — Capsule Opacification; Pseudophakia; Cataract | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Tecnis ZCB00 (Other): eyes with implantation of Tecnis ZCB00
  Interventions: Procedure: intraocular lens implantation
- Acrysof SA60AT (Other): eyes with implantation of Acrysof SA60AT
  Interventions: Procedure: intraocular lens implantation

INTERVENTIONS:
Procedure: intraocular lens implantation

SUMMARY:
Age-related cataract is the main cause of impaired vision in the elderly population worldwide. In the UK, more than half of people who are over 65 have some cataract development in one or both eyes. The only treatment that can restore functional visual ability is cataract surgery where the opacified crystalline lens is removed by phacoemulsification and an artificial intraocular lens is implanted. It is estimated that around 10 million cataract operations are performed around the world each year. Cataract operations are generally very successful, with a low risk of serious complications. The most common risk is developing a condition called posterior capsule opacification (PCO), which causes impaired vision to return.

During the past two decades, cataract surgery underwent tremendous change and modernisation resulting in today's small incision phacoemulsification surgery and a safe technique with a short rehabilitation time for the patient. The most frequent long-term complication of cataract surgery remains to be posterior capsule opacification (PCO). In the past few years, refinements in surgical technique and modifications in IOL design and material have led to a decrease in the incidence of PCO.

It has been shown that a sharp posterior optic edge inhibits migration of lens epithelial cells (LEC) behind the IOL optic and therefore have a lower incidence of posterior capsule opacification (PCO). Most IOL designs have open-loop haptics that are connected to the optic towards the end of the production process, also called multipiece designs.

For several reasons such as better ease of use with injector systems and higher efficiency in the production process, companies have developed IOLs with open-loop haptics out of one block of material, also called single-piece designs. In the case of such single-piece IOLs, the haptics tend to be much thicker than with multipiece IOLs. A potential drawback of the thick haptics maybe an incomplete closure of the capsule at the optic rim with a reduced bending effect of the posterior capsule around the posterior optic edge. Additionally, the posterior sharp edge is often discontinuous in the region of the haptic-optic junctions. These locations may serve as a scaffold for LECs to migrate behind the IOL optic resulting in PCO. Nowadays a multitude of different single piece IOLS are available, many of them similar but of course with some differences in regard to the chemical composition of the acrylic material and the IOL design.

The purpose of this study is to compare the intensity of posterior capsule opacification (PCO) between two different 1-piece foldable hydrophobic acrylic intraocular lenses (IOLs) with different design of the sharp posterior edge within a follow up period of three years.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract
* Good overall physical constitution

Exclusion Criteria:

* History of ocular disease or intraocular surgery
* Laser treatment
* Diabetes requiring medical control
* Glaucoma
* Severe retinal pathology that would make a postoperative visual acuity of 20/40 (decimal equivalent = 0.5) or better unlikely

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Posterior capsule opacification (PCO) | 3 years
  PCO = migration of lens epithelial cells behind the IOL optic after cataract surgery

SECONDARY OUTCOMES:
frequency of neodymium:yttrium-aluminium-garnet (Nd:YAG) capsulotomy | 3 years
  Treatment of PCO in neodymium:yttrium-aluminium-garnet (Nd:YAG) capsulotomy. The frequency of this treatment will be asseseed in absolute and relative (percentage) values

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria